CLINICAL TRIAL: NCT02649712
Title: Unilateral Stenting Versus Bilateral Stenting for Malignant Hilar Biliary Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: xzxy20160106
Record Dates: First submitted 2016-01-06; First posted 2016-01-07 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Cholangiocarcinoma; Gallbladder Carcinoma; Hepatocellular Carcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Gallbladder Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral stent (Active Comparator): Patients undergo placement of unilateral biliary stent on day 1.
  Interventions: Device: biliary stent
- Bilateral stents (Active Comparator): Patients undergo placement of bilateral biliary stents on day 1.
  Interventions: Device: biliary stent

INTERVENTIONS:
Device: biliary stent — Self-expandable biliary nitinol alloys stent

SUMMARY:
The purpose of this study is to compare the clinical effectiveness and long-term outcomes between patients with malignant hilar biliary obstruction who are treated by unilateral or bilateral stenting.

DETAILED DESCRIPTION:
Malignant hilar biliary obstruction is a common clinical manifestation and it can be caused by cholangiocarcinoma, gallbladder carcinoma, liver cancer, or other metastatic carcinoma. Most patients with malignant hilar biliary obstruction are unresectable at diagnosis. Biliary stenting has been widely used in palliative treatment of malignant hilar biliary obstruction.

Hilar biliary obstruction usually involves the bifurcation of the biliary tract. Some researchers recommended unilateral stenting for malignant hilar biliary obstruction because drainage of 25% of entire liver can achieve the clinical success of biliary drainage. However, some researchers recommended bilateral stenting for malignant hilar biliary obstruction because some researches demonstrated that bilateral stenting can achieve a longer stent patency.In addition, there was no significant difference in post stenting survival between patients who were treated by unilateral or bilateral stenting. Therefore, it remains under debate whether unilateral or bilateral stenting is better in the treatment of malignant hilar biliary obstruction.

The purpose of this study is to compare the clinical effectiveness and long-term outcomes between patients with malignant hilar biliary obstruction who are treated by unilateral or bilateral stenting.

ELIGIBILITY:
Inclusion Criteria:

1. Malignant hilar biliary obstruction;
2. Unresectable cases

Exclusion Criteria:

1. Bismuth I patients;
2. inability to obtain informed consent;
3. Eastern Cooperative Oncology Group performance status of 4;
4. severe dysfunction in other organs.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Stent patency (Stent dysfunction is suspected when the patient experiences recurrence of jaundice) | From the date of randomization until the date of first documented stent dysfunction, assessed up to 10 months
  Stent dysfunction is suspected when the patient experiences recurrence of jaundice.

SECONDARY OUTCOMES:
Overall survival | From the date of randomization until the date of first documented death from any cause, assessed up to 12 months
  From the date of randomization until the date of first documented death from any cause.
Stent dysfunction free-patient survival | From the date of randomization until the date of first documented stent dysfunction or the date of death from any cause, whichever came first, assessed up to 10 months.
  From the date of randomization until the date of first documented stent dysfunction or the date of death from any cause, whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Cao, MD, Principal Investigator — Xuzhou Central Hospital
Locations (1):
- Xuzhou Central Hospital, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.

REFERENCES:
- [Background] Iwano H, Ryozawa S, Ishigaki N, Taba K, Senyo M, Yoshida K, Sakaida I. Unilateral versus bilateral drainage using self-expandable metallic stent for unresectable hilar biliary obstruction. Dig Endosc. 2011 Jan;23(1):43-8. doi: 10.1111/j.1443-1661.2010.01036.x. Epub 2010 Nov 30. PMID 21198916
- [Background] Yasuda I, Mukai T, Moriwaki H. Unilateral versus bilateral endoscopic biliary stenting for malignant hilar biliary strictures. Dig Endosc. 2013 May;25 Suppl 2:81-5. doi: 10.1111/den.12060. PMID 23617655
- [Background] Liberato MJ, Canena JM. Endoscopic stenting for hilar cholangiocarcinoma: efficacy of unilateral and bilateral placement of plastic and metal stents in a retrospective review of 480 patients. BMC Gastroenterol. 2012 Aug 9;12:103. doi: 10.1186/1471-230X-12-103. PMID 22873816
- [Background] Gwon DI, Ko GY, Sung KB, Yoon HK, Shin JH, Hyoung Kim J, Kim J, Oh JY. Percutaneous biliary metallic stent placement in patients with unilobar portal vein occlusion caused by advanced hilar malignancy: outcome of unilateral versus bilateral stenting. AJR Am J Roentgenol. 2011 Oct;197(4):795-801. doi: 10.2214/AJR.11.6424. PMID 21940566
- [Background] Mukai T, Yasuda I, Nakashima M, Doi S, Iwashita T, Iwata K, Kato T, Tomita E, Moriwaki H. Metallic stents are more efficacious than plastic stents in unresectable malignant hilar biliary strictures: a randomized controlled trial. J Hepatobiliary Pancreat Sci. 2013 Feb;20(2):214-22. doi: 10.1007/s00534-012-0508-8. PMID 22415652
- [Background] Bulajic M, Panic N, Radunovic M, Scepanovic R, Perunovic R, Stevanovic P, Ille T, Zilli M, Bulajic M. Clinical outcome in patients with hilar malignant strictures type II Bismuth-Corlette treated by minimally invasive unilateral versus bilateral endoscopic biliary drainage. Hepatobiliary Pancreat Dis Int. 2012 Apr;11(2):209-14. doi: 10.1016/s1499-3872(12)60150-7. PMID 22484591
- [Background] Inal M, Akgul E, Aksungur E, Seydaoglu G. Percutaneous placement of biliary metallic stents in patients with malignant hilar obstruction: unilobar versus bilobar drainage. J Vasc Interv Radiol. 2003 Nov;14(11):1409-16. doi: 10.1097/01.rvi.0000096762.74047.a6. PMID 14605106
- [Background] Naitoh I, Ohara H, Nakazawa T, Ando T, Hayashi K, Okumura F, Okayama Y, Sano H, Kitajima Y, Hirai M, Ban T, Miyabe K, Ueno K, Yamashita H, Joh T. Unilateral versus bilateral endoscopic metal stenting for malignant hilar biliary obstruction. J Gastroenterol Hepatol. 2009 Apr;24(4):552-7. doi: 10.1111/j.1440-1746.2008.05750.x. Epub 2009 Feb 12. PMID 19220678
- [Background] Li M, Wu W, Yin Z, Han G. [Unilateral versus bilateral biliary drainage for malignant hilar obstruction: a systematic review and meta-analysis]. Zhonghua Gan Zang Bing Za Zhi. 2015 Feb;23(2):118-23. doi: 10.3760/cma.j.issn.1007-3418.2015.02.009. Chinese. PMID 25880978
- [Derived] Fu YF, Zhou WJ, Shi YB, Cao W, Cao C. Percutaneous stenting for malignant hilar biliary obstruction: a randomized controlled trial of unilateral versus bilateral stenting. Abdom Radiol (NY). 2019 Aug;44(8):2900-2908. doi: 10.1007/s00261-019-02010-6. PMID 30968181